CLINICAL TRIAL: NCT05359822
Title: Investigating the Impact of a Patient-directed Coronary Artery Calcium Score Report: A Randomized-controlled Trial
Brief Title: Investigating the Impact of a Patient-directed Coronary Artery Calcium Score Report
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Sanjay Rajagopalan, Assistant Professor of Medicine and Radiology, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20210601
Record Dates: First submitted 2022-04-28; First posted 2022-05-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Computed Tomography for Calicum Scoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical Standard Report Only (No Intervention): Participants referred for Coronary Artery Calcium Score Test that receive clinical standard CAC risk report only.
- Clinical Standard Report plus Image-Based Report (Experimental): Participants referred for Coronary Artery Calcium Score Test that receive clinical standard CAC risk report plus additional image-based report.
  Interventions: Other: Image-Based Report

INTERVENTIONS:
Other: Image-Based Report — Participants will receive the new coronary artery calcium score risk report plus the old report
  Arms: Clinical Standard Report plus Image-Based Report

SUMMARY:
The goal of this study is to examine if communication of image-based cardiovascular risk to patients undergoing coronary artery calcium scoring (CAC) improves patient understanding of their risk for cardiovascular disease when compared with usual care (physician-only report).

ELIGIBILITY:
Inclusion Criteria:

* Age range: from 40 to 89
* Referred for CAC at UHHS

Exclusion Criteria:

* Less than 40 years of age or over 89 years old.
* Underwent CAC at other locations besides UHHS.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in LDL Cholesterol | baseline-12 months
  Change in LDL cholesterol levels obtained from EMR between baseline to 12 months

SECONDARY OUTCOMES:
Change in Total Cholesterol | baseline-12 months
  Change in Total Cholesterol
Change in Triglycerides | baseline-12 months
  Change in Triglycerides
Change in HDL cholesterol | baseline-12 months
  Change in HDL cholesterol
Change in Weight | baseline-12 months
  Change in Weight
Change in Systolic blood pressure | baseline-12 months
  Change in Systolic blood pressure
Change in Diastolic blood pressure | baseline-12 months
  Change in Diastolic blood pressure
Change in HbA1c | baseline-12 months
  Change in HbA1c
Smoking Cessation Visits as measured by medical record review - yes/no | 12 months
  Smoking Cessation Encounters
Statin prescriptions written as measured by medical record review - yes/no | 12 months
  Statin prescriptions
Aspirin prescriptions written as measured by medical record review - yes/no | 12 months
  Aspirin prescriptions
Stress tests ordered as measured by medical record review - yes/no | 12 months
  Stress testing

OTHER OUTCOMES:
Exploratory: Change in Perception of Risk of Heart Diseases as measured by Perception of Heart Disease Risk score | Baseline, 3 months, 12 months
  Perception of Heart Disease Risk Disease Risk score
Exploratory: Change in Motivation to Change Behavior as measured by Motivation to Change Behavior (TSRQ) Survey Behavior | Baseline, 3 months, 12 months
  Motivation to Change Behavior (TSRQ) Disease Risk score
Exploratory: Change in Medication adherence as measured by Medication adherence (MARSS) Survey | Baseline, 3 months, 12 months
  Changes in medication adherence (MARSS)

CONTACTS AND LOCATIONS:
Overall Officials: Sadeer Al-Kindi, MD, Principal Investigator — University Hospitals

IPD SHARING:
Plan to Share IPD: No